CLINICAL TRIAL: NCT07315529
Title: Legume Consumption Within a Mediterranean Diet Framework and Its Effects on Cellular Hydration, Autonomic Regulation, and Functional Performance in Competitive Swimmers: A Five-Month Intervention Study
Brief Title: Legume-Enriched Mediterranean Diet and Cellular Hydration in Competitive Swimmers
Acronym: LEGUMES-SWIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Raffaele Telematic University (Other)
Responsible Party: Principal Investigator, Mauro Lombardo, Full Professor, San Raffaele Telematic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LEGUMES-SWIM; Lazio Area 5, N.57/SR/23 (Other: Lazio Area 5 Territorial Ethics Committee, Italy)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diet Habits; Athlete
Keywords: Mediterranean diet; Legume consumption; Competitive swimmers; Athletes; Bioelectrical impedance analysis; Phase angle; Extracellular water; Intracellular water; Heart rate variability; Critical swim speed
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Parallel-group interventional study with three diet-based arms: control group with no change in legume intake, moderate-intake group increasing to 3 servings/week, and high-intake group increasing to 6 servings/week, under standardized training conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3-Legumes (Experimental): Competitive swimmers increasing legume intake to 3 servings per week while maintaining usual diet and training load.
  Interventions: Other: Legume-enriched Mediterranean diet
- 6-Legumes (Experimental): Competitive swimmers increasing legume intake to 6 servings per week while maintaining usual diet and training load.
  Interventions: Other: Legume-enriched Mediterranean diet
- Control (No Intervention): Competitive swimmers with habitual legume intake <1 serving/week, receiving no prescribed change in legume consumption.

INTERVENTIONS:
Other: Legume-enriched Mediterranean diet — Adjustment of habitual legume intake within a Mediterranean diet pattern to 3 or 6 servings per week, without altering other dietary components or training regimen.
  Arms: 3-Legumes; 6-Legumes

SUMMARY:
This study investigates whether increasing legume consumption within a Mediterranean diet framework improves cellular hydration, autonomic regulation, and functional performance in competitive swimmers. Thirty-nine adolescent and young adult swimmers were monitored over a five-month competitive season under standardized training conditions. Participants were allocated to three groups according to habitual legume intake: a control group (<1 serving/week, no dietary change), a moderate-intake group (≈2 servings/week increased to 3/week), and a high-intake group (≈3-4 servings/week increased to 6/week). Dietary counseling focused exclusively on adjusting legume intake, while overall training load and other dietary components were maintained. Primary outcomes include bioelectrical impedance-derived phase angle and body water distribution indices (extracellular water, intracellular water, ECW/ICW ratio) as markers of cellular health and hydration. Secondary outcomes include heart rate variability, cardiac coherence as indices of autonomic balance, and critical swim speed as a performance-related measure. The study aims to clarify whether a simple, sustainable increase in legume intake can support athletes' cellular integrity, autonomic function, and functional status without altering standard training programs.

DETAILED DESCRIPTION:
This interventional study was conducted in competitive swimmers to evaluate the impact of higher legume consumption, within a Mediterranean diet framework, on markers of cellular health, body water distribution, autonomic regulation, and functional performance. Thirty-nine competitive swimmers (mean age approximately 20 years; both males and females) were enrolled and followed for five months during the first half of the competitive season. All athletes trained under similar standardized conditions, completing six weekly sessions that combined dry-land pre-activation, in-water training, and, in some sessions, gym-based strength work.

At baseline, participants completed an online dietary assessment using the validated MEDI-LITE questionnaire to quantify adherence to the Mediterranean diet and habitual legume intake. Based on baseline legume consumption, swimmers were assigned to one of three groups: a control group (<1 serving/week, no change in diet), a moderate-intake group (≈2 servings/week increased to 3 servings/week), and a high-intake group (≈3-4 servings/week increased to 6 servings/week). A qualified nutrition professional provided counseling to adjust only legume intake, while other aspects of diet were kept stable. Dietary adherence and legume consumption were monitored regularly throughout the study, and the MEDI-LITE questionnaire was repeated at the end of the intervention.

The primary endpoints are phase angle and hydration indices derived from bioelectrical impedance analysis, including extracellular water (ECW), intracellular water (ICW), and the ECW/ICW ratio, which are considered integrated markers of cellular integrity, cell mass, and fluid compartmentalization. Secondary endpoints include measures of autonomic function-heart rate variability and cardiac coherence-assessed with a standardized device, and a critical swim speed test performed in an indoor pool as a functional performance indicator. Anthropometric data and basic clinical information were also collected.

The study was approved by the Lazio Area 5 Territorial Ethics Committee (Approval Code: N.57/SR/23) and conducted in accordance with the Declaration of Helsinki; all participants provided written informed consent before enrollment. By focusing on a feasible dietary modification (greater legume intake) within an otherwise stable Mediterranean-style eating pattern and unchanged training load, the study is designed to generate sport-specific evidence on whether plant-based protein sources such as legumes can enhance cellular hydration, autonomic regulation, and performance-related parameters in competitive athletes.

ELIGIBILITY:
Inclusion Criteria:

* Competitive swimmers training at least six sessions per week.
* Age ≥18 years.
* Ability to complete an online questionnaire in Italian prior to the first clinical evaluation.
* Willingness to comply with the prescribed legume intake pattern for the assigned group.
* Provision of written informed consent.

Exclusion Criteria:

* Current use of performance-enhancing drugs or any chronic medication.
* Musculoskeletal injury or medical conditions that could interfere with training or study assessments.
* Consumption of alcohol or caffeinated beverages within 15 hours before testing sessions.
* Inability or unwillingness to complete the scheduled assessments or to provide informed consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in phase angle (degrees) | Baseline and 5 months
  Phase angle derived from whole-body bioelectrical impedance analysis, reflecting cellular integrity and body cell mass. Measured at baseline and after 5 months in each arm.

SECONDARY OUTCOMES:
Change in extracellular water percentage (ECW) | Baseline and 5 months
  Extracellular water percentage obtained from bioelectrical impedance analysis, used as an index of fluid distribution.
Change in ECW/ICW ratio | Baseline and 5 months
  Ratio between extracellular and intracellular water derived from bioelectrical impedance analysis, indicating body water compartmentalization.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Open University, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided
At present, there is no finalized institutional policy or dedicated repository for sharing de-identified individual participant data for this study. The investigators may consider data sharing in the future upon development of appropriate governance procedures, data use agreements, and additional ethics committee approvals.